CLINICAL TRIAL: NCT04592081
Title: A Randomized Controlled Clinical Trial aSsessing the Efficacy of DEXTENZA, Sustained Release Dexamethasone 0.4 mg Insert When Placed Within the Upper Eye Lid Canaliculus in Comparison to the Lower Lid Canaliculus Following Bilateral Cataract Extraction Surgery With Posterior Chamber Intraocular Lens Implant (CE/PCIOL).
Brief Title: Dextenza Within Upper Lid Canaliculus Compared With Lower Lid Canaliculus Following Bilateral Cataract Extraction Surgery With PCIOL.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kerry Assil, MD (Other)
Responsible Party: Sponsor-Investigator, Kerry Assil, MD, Sponsor-Investigator, Principal Investigator, Assil Eye Institute
Organization: Assil Eye Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The Assil Study
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Post-Surgical Ocular Pain; Post-Surgical Ocular Inflammation
Keywords: Dexamethasone; Cataract; Capsule Opacification; Inflammation; Lens Diseases; Eye Diseases; Anti-Inflammatory Agents
MeSH Terms: conditions — Cataract; Capsule Opacification; Inflammation; Lens Diseases; Eye Diseases | interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: All patients will receive: First eye randomized for either lower lid (control eye) or upper lid (study eye) insertion and the contralateral eye receiving the opposite site insertion in the OR following CE/PCIOL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEXTENZA placed within the upper canaliculus (Experimental): Dextenza placed within the upper canaliculus following bilateral cataract extraction surgery with posterior chamber intraocular lenses implantation.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- DEXTENZA placed within the lower canaliculus (Active Comparator): Dextenza placed within the lower canaliculus following bilateral cataract extraction surgery with posterior chamber intraocular lenses implantation.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — Dextenza 0.4Mg Ophthalmic Insert

SUMMARY:
Assessing DEXTENZA efficacy when placed within the upper eyelid canaliculus as opposed to the lower eyelid canaliculus.

DETAILED DESCRIPTION:
Randomized controlled clinical trial assessing the efficacy of DEXTENZA, sustained release dexamethasone 0.4 mg insert when placed within the upper eye lid canaliculus in comparison to the lower lid canaliculus following bilateral cataract extraction surgery with posterior chamber intraocular lens implant (CE/PCIOL).

ELIGIBILITY:
Inclusion Criteria:

* Been diagnosed with clinically significant cataract and CE/PCIOL has been planned
* Bilateral cataract surgery with IOL has been planned
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Pregnancy (must be ruled out in women of child-bearing age with pregnancy test)
* Active infectious systemic disease
* Active infectious ocular or extraocular disease
* Obstructed nasolacrimal duct in the study eye(s)
* Hypersensitivity to dexamethasone
* Patients being treated with immunomodulating agents in the study eye(s)
* History of prior ocular surgery, excluding Lasik or PRK
* History of ocular inflammation or macular edema
* Use of any systemic NSAIDs greater than 375 mg per day
* Patients being treated with immunosuppressants and/or oral steroids
* Patients with a corticosteroid implant (i.e. Ozurdex)
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-11 (Estimated)

PRIMARY OUTCOMES:
Post-operative inflammation scores | Assessed on Days 1, 7, 30 for change
  As measured on a scale of 0-4: absence of cell to be defined as a grade of 0-0.5, absence of flare to be defined as a grade of 0-1.
Post-op pain scores | Assessed on Days 1, 7, 30 for change
  As measured on a scale from 0-10

SECONDARY OUTCOMES:
Ease of Insertion (successful implantation) | Assessed on Day 0 (Day of Insertion)
  As measured by Physician Ease of Use Questionnaire
Intraocular Pressure | Assessed on Days 1, 7, 30, 90 for change
  As measured by Goldmann Applanation
Visual Outcome | Assessed at all time points;comparison of Day 30 vs Day 90
  As measured by BCVA
Absence of CME | Assessed on Day -30 to -1 and Day 90 for change
  As measured by OCT
Need of additional steroids | Assessed on Days 1, 7, 30, 90 for change
  As measured by rescue medication added
Absence of rebound iritis | Assessed on Days 1, 7, 30, 90 for change
  As measured by presence of cells
Patient reported outcomes | Assessed on Day 90
  As measured by patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Assil, MD, Principal Investigator — Assil Eye Institute
Locations (1):
- Assil Eye Institute, Beverly Hills, California, United States